CLINICAL TRIAL: NCT07103278
Title: An Open-label, Randomized, Single-dose, 2-sequence, 2-period, Crossover Study to Evaluate the Safety and the Pharmacokinetics of AD-116 Compared to AD-1161 in Healthy Adult Male Volunteers Under Fasting Conditions
Brief Title: A Clinical Trial to Evaluate the Safety and the Pharmacokinetics of AD-116 Compared to AD-1161 in Healthy Adult Male Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-116BE
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1 : Reference Drug(AD-1161), Period 2 : Test Drug(AD-116)
  Interventions: Drug: AD-116; Drug: AD-1161
- Sequence B (Experimental): Period 1 : Test Drug(AD-116), Period 2 : Reference Drug(AD-1161)
  Interventions: Drug: AD-116; Drug: AD-1161

INTERVENTIONS:
Drug: AD-116 — AD-116 Oral Tablet
Drug: AD-1161 — AD-1161 Oral Capsule

SUMMARY:
The study compare and evaluate the safety and pharmacokinetic characteristics between the administration of AD-116 and the administration of AD-1161 in healthy adult male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Body weight equal to or greater than 50kg and Body mass index (BMI) between 18.0 kg/m2 and 30.0 kg/m2 at the time of screening visit
* The Age equal to or greater than 19 in healthy adult male volunteers at the time of screening visit

Exclusion Criteria:

* Participation in another clinical study with an investigational drug within the 6 months from scheduled first administration
* Other exclusions applied

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve during dosing interval (AUCt) | pre-dose (0hour) to 72hours
  AUCt of AD-116
Maximum concentration of drug in plasma (Cmax) | pre-dose (0hour) to 72hours
  Cmax of AD-116

IPD SHARING:
Plan to Share IPD: No